CLINICAL TRIAL: NCT06251531
Title: The Effect of Goal-Directed Therapist-Guided Play-Based Intervention in Children With Cerebral Palsy: A Randomized Controlled Study
Brief Title: Goal-Directed Therapist-Guided Play-Based Intervention in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruya Gul Temel (Other)
Responsible Party: Sponsor-Investigator, Ruya Gul Temel, Occupational Therapist, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ergo.21269652
Record Dates: First submitted 2023-12-06; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Cerebral Palsy
Keywords: play, child, intervention
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GD-TG-PBI (Experimental): Goal-Directed Therapist-Guided Play-Based Intervention
  Interventions: Other: Goal-Directed Therapist-Guided Play-Based Intervention (GD-TG-PBI)
- Control Group (No Intervention): Routine therapy

INTERVENTIONS:
Other: Goal-Directed Therapist-Guided Play-Based Intervention (GD-TG-PBI) — The GD-TG-PBI used play to improve performance in targeted functional activities. The program was planned by a physiotherapist with 25 years' experience and an occupational therapist with six years' experience in play. The sessions were based on motor-learning principles supporting cortical plasticity. Individual-specific goals were transformed into play activities that increase occupational participation with regard to the child's abilities, needs, and learning potential. A top-down approach based on direct gamification was adapted without dividing it into components, instead of a component-based, bottom-up approach. Thus, a structured play program was created and an individual-specific intervention was applied in line with the occupational goals and detailed motor evaluations. Positive, active experiences facilitated the adaptation of the learned skills to daily life.
  Other Names: Goal-Directed Therapist-Guided Play-Based Intervention
  Arms: GD-TG-PBI

SUMMARY:
Abstract Objective: This study planned to examine the effect of Goal-Directed Therapist-Guided Play-Based Intervention (GD-TG-PBI) on occupational performance, occupational satisfaction and functional performance in children with diplegic cerebral palsy (DCP).

Materials and Methods: This study was designed as a randomized controlled trial. 34 children with DCP (14 boys; 20 girls) who received routine therapy included to the study. All children were classified according to the Gross Motor Function Classification System (GMFCS) and the Manual Abilities Classification System (MACS). Participants were randomly divided into two groups: the GD-TG-PBI group (number =17; mean age: 7.70±2.25 years) and the control group (number =17; mean age: 7.41±2.06 years). Both groups received routine therapy twice a week for 45 minutes per session during 8 weeks; while the GD-TG-PBI group received GD-TG-PBI additional to routine therapy twice a week for 45 minutes per session during 8 weeks. Occupational performance and satisfaction were determined with the Canadian Occupational Performance Measure (COPM), and functional performance was evaluated with the Pediatric Evaluation of Disability Inventory (PEDI). The COPM and PEDI were performed before and after the intervention for both groups. Dİfferences between COPM and PEDI values before and after the intervention calculated, additionally the effect size of each parameter calculated.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria of the study were a spastic DCP diagnosis, being aged 4-12 years, Gross Motor Function Classification System (GMFCS) level I, II or III, and Manual Ability Classification System (MACS) level I or II, and ability to follow verbal instructions.

Exclusion Criteria:

* The exclusion criteria were mental retardation diagnosis, additional treatment other than neurodevelopmental treatment (NDT), surgical intervention or Botulinum Toxin injection in the last six months, diagnosis of psychiatric disorder accompanying CP, vision and/or hearing problems affecting participation.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
The Canadian Occupational Performance Measure (COPM) | 30 minutes
  It was used to identify children's occupational problems and determine the goals of play. The COPM is a patient-reported, semi-structured assessment for individuals aged 8 years and over; it is used for goal-setting and planning interventions (18). The participants who were older than 8 years were asked to answer by themselves, and participants who were under 8 years answered both by themselves and parent proxy to identify and score occupational performance problems experienced in self-care, productivity, and leisure. In comparing initial and final values, a change of at least 2 points indicates clinical significance (19,20). The Turkish validity and reliability was established by Torpil et al (20).
Pediatric Evaluation of Disability Inventory (PEDI) | 30 minutes
  It was used to evaluate functional performance and disability level.PEDI contains 3 scales : Functional Skills Scale (FSS) that identifies clinical patterns of current skills in functional skill attainment; Caregiver Assistance Scale that indirectly measures capability and evaluates actual performance by assesing the extent of help a parent provides in daily functioning, and Modifications scale which was not used in current study. The FSS consists of self-care, mobility, and social function, including the ICF's activity and participation. It consist 197 items in total devided as 73 items in self care, 59 items in mobility and 65 items in social function. Each item is scored as unable (0) or able (1). The caregiver assistance scale measures the caregiver support with a Likert-type rating (0-5). PEDI is sensitive to show clinical changes that can guide the therapist in defining the functional level of children with CP (21-22). The Turkish validity and reliability was established (22).
Gross Motor Function Classification System (GMFCS) | 15 minutes
  The GMFCS was used for classify motor functions of participants. The GMFCS consisted five levels from 1 to 5, level 1 is the most independent whereas level 5 is fuly dependent. The Turkish GMFCS is valid and reliable.
Manual Ability Classification System (MACS) | 15 minutes
  The MACS was used for classify manuel functions of participants. The MACS consisted five levels from 1 to 5, level 1 is the most independent whereas level 5 is fuly dependent. The Turkish MACS is valid and reliable.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Rüya Gül Temel, Ankara, Etimesgut
  - Rüya Gül Temel, Ankara

IPD SHARING:
Plan to Share IPD: No